CLINICAL TRIAL: NCT04824781
Title: Recovery From Paranoia: a Qualitative Exploration
Status: Completed | Type: Observational
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Other Study IDs: PID 15402; HRA (Other: 21/WA/0081); IRAS (Other: 289951)
Record Dates: First submitted 2021-03-25; First posted 2021-04-01 (Actual); Last update posted 2022-05-19 (Actual); Status verified 2021-03

CONDITIONS: Paranoia; Persecutory Delusion
Keywords: Paranoia; Persecutory delusions; Recovery; NHS; Qualitative; Interpretative phenomenological analysis
MeSH Terms: conditions — Paranoid Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Qualitative interview — Participants will be interviewed about their experiences of recovery from paranoia.

SUMMARY:
Paranoia, the experience of undue or excessive mistrust, exists on a continuum which includes suspicious thoughts, ideas of reference, and persecutory delusions. Persecutory delusions refers to strong unfounded fears that others intend harm. These fears are very common. They affect around 70% of patients with schizophrenia. They can be distressing and make day-to-day tasks difficult. However, current treatments are limited and a significant proportion of people do not benefit sufficiently. Therefore, improvements in treatment are needed. A better understanding of the experience of recovery from paranoia will help inform theoretical understanding and treatment development. Currently we do not fully understand what causes paranoia to occur, persist, or end. As such, it is critical to understand the experiences of those who have recovered, in particular what elements encourage recovery. Therefore, the aim of this study is to gain a first-person perspective on how people recover from paranoia and what psychological processes are important for recovery from paranoia. Using a qualitative approach appropriate for exploratory research, semi-structured interviews will be conducted with 12-15 patients who have recovered from paranoia. Interviews will be analysed using interpretative phenomenological analysis, a qualitative research approach which aims to provide insight on how an individual, in a particular situation, makes sense of their experience.

ELIGIBILITY:
Inclusion Criteria:

* Participant has recovered from the paranoia. This is defined as: A.) conviction in persecution beliefs is rated as less than 10% and B.) not experiencing significant distress related to paranoia and C.) currently scoring outside the clinical range of the revised Green et al., Paranoid Thoughts Scale (R-GPTS; Freeman, 2019);
* Participants should have had experiences of paranoia in the context of non-affective psychosis. This will be determined by participant's agreement that they previously had the sort of thoughts listed in the revised Green et al. Paranoid Thoughts Scale (R-GPTS; Freeman, 2019);
* Participant is currently a patient of Oxford Health NHS Foundation Trust;
* Participant is willing and able to give informed consent for participation in the study;
* Aged 16 years or above;
* Participant has sufficient English language skills to participate in the interview.

Exclusion Criteria:

The following exclusion criteria will apply based on concerns regarding risk and capacity to consent:

* Currently experiencing acute psychiatric symptoms which preclude ability to participate in a sustained interview;
* Diagnosis of a moderate to severe intellectual disability;
* High levels of associated risk to self or to others e.g. actively suicidal;
* Primary diagnosis of alcohol or drug misuse; personality disorder; significant forensic history;
* At the time of recruitment COVID-19 restrictions do not permit face-to-face interviews and the participant is not willing or able to conduct the interview remotely via video call.

Min Age: 16 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: A sample of approximately 15 patients who have recovered from paranoia will be recruited. Participants will be recruited according to the inclusion and exclusion criteria adumbrated below.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2021-06-09 (Actual); Primary Completion 2021-07-27 (Actual); Study Completion 2022-02-16 (Actual)

PRIMARY OUTCOMES:
Qualitative interview accounts | March 2021-March 2022
  Semi-structured interpretative phenomenological analysis (IPA) interviews will be used.

CONTACTS AND LOCATIONS:
Overall Officials: Dr Felicity Waite, DClinPsy, BSc (Hons), Study Director — University of Oxford
Locations (1):
- Oxford Health NHS Foundation Trust, Oxford, Oxfordshire, United Kingdom